CLINICAL TRIAL: NCT04954183
Title: Development of an EEG Diagnostic for Alzheimer's Disease: A Feasibility Study
Brief Title: Development of an EEG Diagnostic for Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Spark Neuro Inc. (Industry)
Responsible Party: Principal Investigator, Erik K. St Louis, Principal Investigator, Mayo Clinic
Other Study IDs: 21-000676
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Dementia With Lewy Bodies; Normal Control APOE e4 Carriers and Noncarriers
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to collect and compare electroencephalogram data from all stages of Alzheimer's disease from preclinical through severe dementia.

DETAILED DESCRIPTION:
Patients with diagnoses of sporadic and late onset Alzheimer's disease dementia, MCI, and DLB evaluated by a dementia subspecialist will meet published diagnostic criteria, and EEGs will be obtained through written informed consent. Regarding presymptomatic patients, we have previously shown that the mean age of MCI diagnosis in our cohort is 73 years and that preclinical cognitive decline begins as much as 20 years before clinical diagnosis but is also affected by APOE genotype. Eligibility therefore will include unimpaired APOE e4/4 homozygotes age 65-75 and APOE e3/4 heterozygotes age 75-85 for the preclinical AD subset and age, sex, and education matched APOE e4 noncarriers for the unaffected controls. Biomarker confirmation for preclinical diagnosis will be utilized to the extent possible (a subset of 130 members of our cohort have undergone amyloid-PET resulting in approximately 45 who are amyloid positive). EEG data will be performed during wakefulness with 15 minutes of eyes open and 15 minutes of eyes closed. A 32 electrode cap will be applied following the 10-20 anatomical system by certified EEG technologists. Data will be recorded using a research-grade EEG system with FDA 510(k) clearance for use in medical contexts. Subjects will be seated in a testing room with minimal distractions. An EEG tech will fit the subject with a cap containing NN Ag/AgCl electrodes placed according to the international 10-10 system and ensure electrode impedances stay below 10 kΩ. Subjects will be instructed to minimize movements and remain in a relaxed but wakeful state. We will record fifteen minutes of eyes-open resting state EEG. Afterwards, the subjects will be instructed to close their eyes and reminded to stay relaxed but awake, and we will record fifteen minutes of eyes-closed resting state EEG. During the recording session, a researcher will monitor the subject's behavior and the EEG signal. The researcher will briefly prompt the subject to remain awake if the subject's behavior or EEG traces show signs of drowsiness. All data will be de-identified then transferred to SPARK Neuro's research and development team for analysis via secure encrypted methods. The data will be stored on password-protected computer systems, and only the necessary research and research-support staff at SPARK Neuro will have access to the data. The SPARK Neuro research and development team will analyze de-identified patient data to address the aims of this proposal. SPARK Neuro will use various techniques including those standard in EEG analysis (e.g. filtering, scaling, independent components analysis), particular approaches shown to be successful in the Alzheimer's disease EEG classification literature (e.g. coherence, relative power in standard frequency bands, functional connectivity, spectral entropy), as well as approaches from the broader machine-learning and EEG literature (e.g. spectral clustering, convolutional neural networks, cross-frequency coupling, non-linear kernels, Katz fractal dimension, beamforming).

ELIGIBILITY:
Inclusion Criteria:

* 5 individuals with moderate to severe dementia, 5 with mild stage dementia, 5 with amnestic MCI, 5 presymptomatic APOE e4 carriers, and 5 age, sex, and education matched APOE e4 noncarriers. Additionally we will include a group of 5 patients with mild to moderate stage dementia with Lewy bodies (DLB), the second most common degenerative dementia, to explore differences from clinically typical Alzheimer's disease patients given the known clinical differences in EEG dysrhythmic severity between them (total of 30).
* Unimpaired APOE e4/4 homozygotes age 65-75 and APOE e3/4 heterozygotes age 75-85 for the preclinical AD subset and age, sex, and education matched APOE e4 noncarriers for the unaffected controls.
* Biomarker confirmation for preclinical diagnosis will be utilized to the extent possible (a subset of 130 members of our cohort have undergone amyloid-PET resulting in approximately 45 who are amyloid positive).

Exclusion Criteria:

* Previous stroke.
* Severe head injury.
* Craniotomy.
* Any other potentially confounding neurologic illness (typically anything that causes structural brain damage).
* Psychoactive medication use will not be an absolute exclusionary criterion in patients with moderate to severe dementia but patients who are relatively drug-free will be prioritized to the extent they are available within the study period.
* Psychoactive drug use will be exclusionary in the prospectively obtained clinical patients.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with moderate to severe dementia, mild stage dementia, amnestic MCI, presymptomatic APOE e4 carriers, and age, sex, and education matched APOE e4 noncarriers will be recruited at Mayo Clinic Arizona to obtain EEG data.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Obtain electroencephalogram (EEG) data | 1 year
  Number of EEG data on individuals at all stages of Alzheimer's disease from preclinical through severe dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Erik K. St. Louis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No